CLINICAL TRIAL: NCT05976906
Title: A Study to Evaluate the Safety, Tolerability, Preliminary Efficacy, Pharmacodynamics and Immunogenicity of Universal CNK-UT Cells in Patients With Advanced Solid Tumors.
Brief Title: Universal Dual-target NKG2D-NKp44 CAR-T Cells in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, Director, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNK-UT-IIT202201
Record Dates: First submitted 2023-05-10; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CNK-UT cells therapy (Experimental): 1. Dose Escalation： Cohort A：Intravenous injection of CNK-UT cells directly. Cohort B：Intravenous injection of CNK-UT cells after preconditioning by fludarabine and cyclophosphamide.
  2. Indications Expansion:
  Intravenous injection of CNK-UT cells according to the results of dose escalation.
  Interventions: Biological: Universal Chimeric Natural Killer Receptor Modified T-cells (CNK-UT)

INTERVENTIONS:
Biological: Universal Chimeric Natural Killer Receptor Modified T-cells (CNK-UT) — 1. Dose Escalation: After enrollment, participants will recieve preconditioning by lymphodepletion or not, and then will be treated with CNK-UT cells with a "3 +3" design to determine the maximum tolerated dose. 3 dose level of CNK-UK cells will be tested: 4.6E6/kg，1.5E7/kg，4.6E7/kg. The participants will first receive a single ascending dose(SAD) mode of administration. During the DLT observation period (21 days), if the participants do not experience DLT, they will receive a multiple ascending dose(MAD) mode of administration.
  2. Indications Expansion: It will be carried out after all participants have completed the DLT observation in the Dose Escalation phase. The target population, dosage and frequency of drug administration in the indication expansion stage can be adjusted and determined according to the previous research results.

SUMMARY:
This is a single arm, open-label, multi-center, phase I study to evaluate the safety, tolerability, preliminary efficacy, pharmacodynamics and immunogenicity of universal chimeric natural killer receptor modified T-cells (CNK-UT) targeting NKG2D-Ligands and NCR2-Ligands with or without lymphodepletion in advanced solid tumors.

DETAILED DESCRIPTION:
This is a single arm, open-label, multi-center, phase I, dose escalation/indications expansion study to assess the safety and tolerability of CNK-UT cells therapy, and to obtain the preliminary efficacy, pharmacodynamics and immunogenicity result in participants who have been diagnosed with advanced solid tumors and failed to standard systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years (including 18 and 70 years old), male or female;
2. Participants with advanced solid tumor diagnosed by histology or cytology (or patients with clinically diagnosed hepatocellular carcinoma) have recurrence or disease progression after first or second-line treatment (with metastasis not excluded). Either the existing standard regimen has failed or cannot be tolerated, or the researchers believe that the participants are not suitable for standard treatment for medical reasons (The Dose Escalation Stage is not limited to the types of tumors, including but not limited to advanced hepatocellular carcinoma, advanced colorectal cancer, advanced cholangiocarcinoma, advanced renal cell carcinoma, advanced triple negative breast cancer, melanoma, sarcoma etc. The Indications Expansion Stages include advanced hepatocellular carcinoma, advanced colorectal cancer, advanced cholangiocarcinoma, advanced renal cell carcinoma, advanced triple negative breast cancer, melanoma, sarcoma).
3. According to the RECIST 1.1, there is at least one measurable target lesion, or a measurable lesion with definite progression after local treatment (based on RECIST v1.1 standard);
4. ECOG physical status score 0 or 1;
5. Estimated life expectancy > 12 weeks;
6. Adequate organ and bone marrow function, and the laboratory test value meets the following requirements within 7 days before enrollment, as follows:

   Blood Routine Test: Absolute neutrophil count (ANC)≥1.0×10^9/L; Platelet count ≥75×10^9/L; Haemoglobin≥9.0 g/dL; Hepatic function：Total bilirubin≤3×ULN; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT)≤5×ULN; Serum albumin≥28 g/L; Renal function: Serum creatinine≤1.5×ULN, or Creatinine clearance rate (CCR)≥60 mL/min (Cockroft-Gault formula); Coagulation function: International normalized ratio (INR)≤1.5×ULN.
7. All toxic responses originating from previous radiotherapy, chemotherapy, or other treatments (occurring within 4 weeks or 5 half-lives of anti-tumor drugs therapy [including but not limited to chemotherapy, targeted therapy, immunotherapy, Chinese herbal medicine]) have returned to NCI CTCAEV5.0 Grade≤1 (except for hair loss);
8. Sufficient venous access for intravenous infusion or venous blood collection;
9. Female participants of childbearing age must undergo a serum or urine pregnancy test before enrollment, and the results must be negative, and agree to take acceptable measures to minimize the possibility of pregnancy during the trial; For female participants of childbearing age or male participants whose sexual partners are women of childbearing age, effective contraceptive measures should be taken during the study and for at least 6 months following the last dose of the study cells infusion.
10. participants voluntarily participate in clinical trial; Understand and know this study, sign an informed consent form, and be willing to follow all experimental procedures.

Exclusion Criteria:

1. Suffering from other malignant tumors or diagnosed within 5 years before enrollment, excluding radical skin basal cell carcinoma, skin squamous cell carcinoma, thyroid cancer, breast cancer (ductal carcinoma in situ) and / or radical resection of carcinoma in situ.
2. Participants with a history of organ transplantation;
3. Participants with symptomatic central nervous system (CNS) metastasis confirmed by imaging or pathological examination and clinically unstable for at least 14 days prior to randomization who require steroid treatment.
4. Presence of gastroesophageal variceal hemorrhage caused by portal hypertension in the past 3 months; evidence of portal hypertension, assessed by researchers as having a high risk of bleeding.
5. Presence of any life-threatening bleeding occurred in the past 3 months, including the need for blood transfusion, surgery or local treatment, and continuous drug treatment.
6. Presence of arterial and venous thromboembolism events in the past 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis or any other serious thromboembolism history. Except for implantable intravenous infusion port or catheter-derived thrombosis, or superficial venous thrombosis, thrombus stability after routine anticoagulant therapy.Allow prophylactic use of small doses of low molecular weight heparin (such as enoxaparin 40 mg/day).
7. Severe bleeding tendency or coagulation dysfunction, or undergoing thrombolytic therapy.
8. Uncontrollable hypertension, systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg after optimal medical treatment, history of hypertensive crisis or hypertensive encephalopathy.
9. Symptomatic congestive heart failure (New York Heart Association Class II-IV). Symptomatic or poorly controlled arrhythmia. History of congenital long QT syndrome or corrected QTc > 500ms during screening (calculated by Fridericia method).
10. Participants with pulmonary diseases such as pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, severe lung function impairment, and Participants with COVID-19 and severe lung function damage caused by viral infection.
11. Active pulmonary tuberculosis (TB), who is receiving anti-tuberculosis treatment or has received anti-tuberculosis treatment within 1 year before enrollment; human immunodeficiency virus (HIV) infection, known syphilis infection.
12. Severe infections that are active or poorly controlled clinically. Severe infection within 4 weeks prior to the initiation of the study, including but not limited to hospitalization due to infection, bacteremia, or complications of severe pneumonia.
13. Active autoimmune diseases that require systemic treatment (such as the use of disease relieving drugs, corticosteroids, or immunosuppressants) have occurred within 2 years prior to the initiation of the study. Allowing the use of alternative therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency), with a known history of primary immunodeficiency. Patients with only positive autoimmune antibodies need to confirm the presence of autoimmune diseases based on the judgment of the investigator.
14. Participants who have received local treatment for advanced tumors within 4 weeks prior to the initiation of the study.
15. Participants who have received radiation therapy within 4 weeks prior to the initiation of the study. For participants who receive radiation therapy 4 weeks before the first administration, all of the following conditions must be met before enrollment: no toxic responses related to radiation therapy, no need to take glucocorticoids, excluding radiation pneumonia, radiation hepatitis, and radiation enteritis; palliative radiotherapy for bone metastases lesion is allowed, which must be completed 2 weeks before enrollment.
16. Participants who have received traditional Chinese medicine with anti-tumor effects or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, except for drugs that need to be used locally to control pleural or ascites) within 2 prior to the initiation of the study.
17. Participants who have received adjuvant surgical therapy, chemotherapy (6 weeks for mitomycin and nitrosourea), targeted therapy, and immunosuppressive therapy 4 weeks prior to the initiation of the study, such as corticosteroid users;
18. Participants who have received treatment from other clinical trials within 12 weeks prior to the initiation of the study.
19. Participants who receive attenuated live vaccines within 6 months prior to the initiation of the study or plan to receive them during the study period.
20. Participants who have undergone major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the initiation of the study, or have severe unhealed wounds, ulcers, or fractures.
21. Uncontrolled/uncorrectable metabolic disorders or other non-malignant organ diseases or systemic diseases or secondary reactions to cancer, which can lead to higher medical risk and/or uncertainty in survival assessments.
22. Allergic to components of CNK-UT injection.
23. Participants suffer from known mental or substance abuse disorders, which may interfere with their ability to comply with research requirements.
24. Women who are pregnant or breastfeeding, as well as male or female participants who have planned for birth within 1 year after receiving medication.
25. Other situations that the participant is identified by the investigator as unsuitable to participate in the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | up to 1 year
  Incidence of Treatment Related AEs, AEs of special interest and serious adverse events (SAEs) assessed by NCI-CTCAE v5.0 criteria
Identification of Maximum Tolerated Dose (MTD) & incidence of Dose-limiting Toxicities (DLTs) | up to 21 days since first infusion of CNK-UT
  Incidence of dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 1 year
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%). In the event of PR or CR, the participants should confirm it no less than 4 weeks after the first evaluation
Disease control rate (DCR) | up to 1 year
  The number of cases in which response are achieved from the start of cells infusion/the total number of evaluable cases (%)
Best overall response(BOR) | up to 1 year
  The best efficacy recorded from the beginning of treatment to the progression or recurrence of the disease
Duration of response (DOR) | up to 1 year
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause
Progression-free survival (PFS) | up to 1 year
  The period from the day when the participant receives the infusion of cellss to the first recorded tumor progression (whether treated or not) or death of any cause, which occurs first
Overall survival (OS) | up to 1 year
  The period from the first infusion to any cause of death
Pharmacokinetics (PK) | up to 48 weeks
  CNK-UT DNA in peripheral blood detected by q-PCR after infusion
Pharmacodynamics (PD) | up to 48 weeks
  IL-2, IFN-γ, TNF-α
tumor marker | up to 48 weeks
  specific tumor related biomarker(such as CEA、CA19-9，CA125、CA50、CA242、AFP) will be analyzed
Immunogenicity | up to 48 weeks
  Antidrug antibodies (ADA) in peripheral blood detected by q-PCR

OTHER OUTCOMES:
biomarkers | Enrollment
  Detection the expression of NKG2D ligand, NKp44 ligand, PD-L1, TIL infiltration ( biomarkers related to clear indications in tumor tissue using immunohistochemical methods, such as RAS and BRAF gene mutations, MSI/MMR, etc. in colorectal cancer.)
HLA typing | Baseline
  Evaluate the impact of HLA typing matching between donors and participants on the survival time and efficacy of CNK-UT in vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Weijia Fang, Principal Investigator — Zhejiang University
Locations (1):
- First affiliated hospital, School of Medicine, Zhejiang University, Hangzhou, China